CLINICAL TRIAL: NCT01913925
Title: Effect of Tyrosine Supplementation on Cognitive Performance and Mood During Military Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H08-05
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Reaction to Severe Stress, Unspecified

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tyrosine-Containing Food Bar (Active Comparator): 150 mg/kg dose of tyrosine per administration, administered twice
  Interventions: Other: Tyrosine-Containing Food Bar
- Placebo bar (Placebo Comparator): 0 mg/kg dose of tyrosine per administration, administered twice
  Interventions: Other: Placebo Bar

INTERVENTIONS:
Other: Tyrosine-Containing Food Bar
  Arms: Tyrosine-Containing Food Bar
Other: Placebo Bar
  Arms: Placebo bar

SUMMARY:
The objective of this research is to determine if tyrosine, an amino acid found in protein-containing foods, will mitigate the cognitive deficits and adverse effects on behavior and mood produced by exposure to military stress. This study was conducted at the US Navy Survive, Evade, Resist, Escape (SERE) school at Brunswick, Maine (ME).

Tyrosine is the dietary precursor of the catecholamine norepinephrine, a key brain neurotransmitter that is critical for the central nervous system (CNS) response to various types of acute stress. Psychological stress increases catecholamine turnover in the brain, increasing the requirement for tyrosine to support synthesis of norepinephrine. Animal and human studies have shown that tyrosine supplementation can produce beneficial effects on cognitive and physiological functions during exposure to a variety of acute stressors.

This project will determine if volunteers treated with supplemental tyrosine during stressful phases of SERE training experience less degradation in cognitive performance and mood than volunteers treated with placebo. Tyrosine or placebo will be administered in a specially developed food bar provided to volunteers. The bar is part of a prototype of ration-component designed for use during assault operations. A between-subjects, double blind experimental design will be employed. Tyrosine, an amino acid found in most protein-containing foods, has been tested in hundreds of volunteers without adverse effects.

Approximately 100 volunteers will be recruited from several SERE classes to ensure up to 80 volunteers complete the study. They will be tested during several portions of SERE. A comprehensive but brief battery of cognitive tests, as well as saliva samples, and heart rate data will be collected in a manner that does not interfere with ongoing training.

Hypotheses:

1. Exposure to the stressors of SERE school will adversely impact cognitive performance and mood of volunteers.
2. The adverse effects of psychological stress on cognitive performance and mood during SERE school will be reduced when volunteers are given supplemental tyrosine compared to placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military enrolled in the US Navy SERE School, Brunswick, ME.
* Fluent in English (non-native English speakers can be enrolled).

Exclusion Criteria:

* None.

[All volunteers enrolled in SERE school require a medical clearance. No additional inclusion or exclusion criteria are necessary.]

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
change from baseline cognitive function compared to cognitive function as measured following treatment administration | baseline and final week of training (approximately 1 week later)

CONTACTS AND LOCATIONS:
Overall Officials: Harris R. Lieberman, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- US Navy SERE School, Brunswick, Maine, United States